CLINICAL TRIAL: NCT01695564
Title: Comparison of Safety and Efficacy of Left Atrial Appendage Occlusion Devices
Brief Title: Safety and Efficacy of Left Atrial Appendage Occlusion Devices
Status: Completed | Type: Observational
Sponsor: Kansas City Heart Rhythm Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 13240
Record Dates: First submitted 2012-07-05; First posted 2012-09-28 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
Keywords: atrial enlargement; left atrial appendage
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- WATCHMAN: Patients that had the WATCHMAN device implanted
  Interventions: Device: WATCHMAN
- LARIAT LAA Device: patients that had LARIAT LAA device implanted
  Interventions: Device: LARIAT LAA

INTERVENTIONS:
Device: LARIAT LAA — The LARIAT snare device is an over-the-wire device guided over the LAA to enable ligation of the LAA. The LARIAT can be opened and closed as desired for ideal positioning without risk of suture deployment.
  Groups: LARIAT LAA Device
Device: WATCHMAN — The WATCHMAN is an expandable device deployed in the LAA via a trans-septal catheter. The implanted device has a self-expanding nitinol frame to secure it in the LAA. The fabric of the WATCHMAN device is permeable to blood.
  Groups: WATCHMAN

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac rhythm disorder in clinical practice. In the last two decades the number of hospitalizations for AF has increased two- to three-fold. More than 6 million people worldwide suffer from atrial fibrillation (AF), a cardiac disorder that results in systemic emboli. Patients with AF are 5 times more likely to have a stroke compared with those without AF.

This registry will collection information on two devices that are used to treat AF. The WATCHMAN and LARIAT. The differences in techniques and subsequent effects of the two devices on outcomes related to AF has not been studied. This study will look to compare the two devices to see how the outcomes may vary.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a LARIAT LAA device occlusion

Exclusion Criteria:

* Patients who have PFO/ASD/critical carotid artery (>70% blockage) disease and hemorrhagic strokes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a LARIAT LAA device occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2012-05; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Effect of LAA occlusion by LARIAT device | Change from Day 0 to Day 90
  This registry will provide data on patient outcomes at different times during follow up. This includes: changes in the appendage size, shape and patients medical history.
Effect of LAA occlusion by LARIAT device | Change from Day 0 to 356 post-procedure
  This registry will provide data on patient outcomes at different times during follow up.This includes: changes in the appendage size, shape and patients medical history.

SECONDARY OUTCOMES:
Compare effectiveness of LAA occlusion procedure by evaluating LAA jet velocities | Days 0, 90, 180, 365 post-procedure and annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States